CLINICAL TRIAL: NCT03342027
Title: Optimizing Smoking Cessation Interventions for People Living With HIV in Nairobi, Kenya
Brief Title: Smoking Cessation Interventions for People Living With HIV in Nairobi, Kenya
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Seth Himelhoch, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: HP-00077523
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: HIV; Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Bupropion

STUDY DESIGN:
Intervention Model Description: 4 conditions: (1) bupropion + Positively Smoke Free (an 8 session tailored behavioral intervention for PLWH smokers); (2) bupropion + Standard of Care (brief advice to quit); (3) Placebo + Positively Smoke Free; and (4) Placebo + Standard of Care.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Bupropion + Positively Smoke Free (Experimental): Positively smoke free-- an 8 session tailored behavioral treatment for smoking cessation bupropion--used for smoking cessation
  Interventions: Drug: Bupropion; Behavioral: Positively smoke free
- Bupropion + Standard of Care (Experimental): Standard of Care--brief advice to quit provided in a standardized format bupropion--used for smoking cessation
  Interventions: Drug: Bupropion; Other: Brief advice to quit smoking
- Placebo + Positively Smoke Free (Experimental): Placebo--matched to bupropion Positively smoke free-- an 8 session tailored behavioral treatment for smoking cessation
  Interventions: Behavioral: Positively smoke free
- Placebo + Standard of Care. (Placebo Comparator): Placebo--matched to bupropion Standard of Care--brief advice to quit provided in a standardized format
  Interventions: Other: Brief advice to quit smoking

INTERVENTIONS:
Drug: Bupropion — medication for smoking cessation
  Other Names: Zyban
  Arms: Bupropion + Positively Smoke Free; Bupropion + Standard of Care
Behavioral: Positively smoke free — an 8 session, tailored behavioral intervention for treating tobacco dependence
  Arms: Bupropion + Positively Smoke Free; Placebo + Positively Smoke Free
Other: Brief advice to quit smoking — Standardized brief advice to quit smoking (standard of care)
  Arms: Bupropion + Standard of Care; Placebo + Standard of Care.

SUMMARY:
The proposed study will use a factorial design to evaluate the most promising and accessible behavioral and pharmacologic treatments aimed at achieving maximal efficacy for smoking cessation among people living with HIV who smoke. The study will randomize 300 participants people living with HIV , who smoke and who are receiving care in HIV clinics affiliated with the Center for International Health, Education, and Biosecurity in Nairobi, Kenya to one of the following 4 conditions: (1) bupropion + Positively Smoke Free (an 8 session tailored behavioral intervention for people living with HIV smokers); (2) bupropion + Standard of Care (brief advice to quit); (3) Placebo + Positively Smoke Free; and (4) Placebo + Standard of Care.

DETAILED DESCRIPTION:
The proposed study will use a factorial design to evaluate the most promising and accessible behavioral and pharmacologic treatments aimed at achieving maximal efficacy for smoking cessation among people living with HIV who smoke. The will randomize 300 participants people living with HIV, who smoke and who are receiving care at HIV clinics affiliated with the Center for International Health, Education, and Biosecurity in Nairobi, Kenya to one of the following 4 conditions: (1) bupropion + Positively Smoke Free (an 8 session tailored behavioral intervention for people living with HIV smokers); (2) bupropion + Standard of Care (brief advice to quit); (3) Placebo + Positively Smoke Free; and (4) Placebo + Standard of Care. The study will use a factorial design as it is a highly efficient method of assessing multiple treatments in a single trial with the possibility of saving both time and resources. All participants will be assessed at baseline,12 weeks and 36 weeks with the main outcome being 7-day abstinence (defined as self-reported no smoking in the past 7 days + CO<7 ppm).

ELIGIBILITY:
Inclusion Criteria

* Chart diagnosis of HIV at recruitment clinic.
* Age 18 years and older
* Currently self-report smoking approximately 1 cigarette per day.
* Motivation to quit (score 6-8 on the Abrams and Briener Readiness to Quit Ladder)
* Able to read and speak English or Swahili
* Willingness and ability to provide informed consent to participate

Exclusion Criteria:

* Has a history of seizure disorder or bulimia nervosa
* Recent use of Bupropion (by participant report in the past 3 months)
* Previous allergic reaction/hypersensitivity to Bupropion (by participant report ever in lifetime)
* Pregnant, nursing, or becoming pregnant during the study (pregnancy test)
* Current use of any medication that would interfere with the protocol in the opinion of a medically accountable Physician
* Known plans to re-locate or travel away from the study site for more than two consecutive months during the study period.
* Expected survival of less than 6 months
* Meets criteria for dementia by scoring below 10 on the Hopkins HIV Dementia Scale.
* The study physician believes that the individual is not medially stable enough to participate in the study. This exclusion will be based on a review of the individual's past medical history and current medical status.
* Based on screening, not meeting criteria for moderate or severe substance disorder as established by the MINI International Neuropsychiatric Interview.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for International Health, Education, and Biosecurity (CIHEB), Kilimani, Nairobi County, Kenya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Keith A, Dong Y, Shuter J, Himelhoch S. Behavioral Interventions for Tobacco Use in HIV-Infected Smokers: A Meta-Analysis. J Acquir Immune Defic Syndr. 2016 Aug 15;72(5):527-33. doi: 10.1097/QAI.0000000000001007. PMID 27028502

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupropion + Positively Smoke Free | Bupropion + Standard of Care | Placebo + Positively Smoke Free | Placebo + Standard of Care.
Started | 74 | 74 | 76 | 76
Completed | 72 | 72 | 74 | 76
Not Completed | 2 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion + Positively Smoke Free | Bupropion + Standard of Care | Placebo + Positively Smoke Free | Placebo + Standard of Care. | Total
Number analyzed (Participants) | 72 | 72 | 74 | 76 | 294
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (10.2) | 40.8 (10.1) | 43.5 (10.2) | 44.2 (10.1) | 42.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 48 | 20 | 56 | 144
  Male | 52 | 24 | 54 | 20 | 150
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 72 | 72 | 73 | 76 | 293
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 72 | 72 | 74 | 76 | 294

OUTCOME MEASURES:

1. Primary Outcome: 7-day Abstinence
Description: defined as self-reported no smoking in the past 7 days + CO<7 ppm
Time Frame: Up to 36 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Bupropion + Positively Smoke Free | Bupropion + Standard of Care | Placebo + Positively Smoke Free | Placebo + Standard of Care.
Number analyzed (Participants) | 72 | 72 | 74 | 76
Participants | 4 | 17 | 15 | 29

ADVERSE EVENTS:
Time Frame: We collected SAEs, All-Cause mortality and Adverse Events from the start of the study until the last participant was completed their final appointment. After a participant completes a baseline, they return 2, 4 and 8 weeks later to review any side effects or concerns from the study medication/placebo. 12- and 36-weeks post baseline, additional interviews are completed to review any new side effects, Adverse Events or SAEs.
Arm/Group | Bupropion + Positively Smoke Free | Bupropion + Standard of Care | Placebo + Positively Smoke Free | Placebo + Standard of Care.
All-Cause Mortality (participants affected / at risk) | 3/72 | 0/72 | 3/74 | 0/76
Serious Adverse Events (participants affected / at risk) | 1/72 | 1/72 | 4/74 | 2/76
Other Adverse Events (participants affected / at risk) | 21/72 | 24/72 | 34/74 | 28/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion + Positively Smoke Free (N=72) | Bupropion + Standard of Care (N=72) | Placebo + Positively Smoke Free (N=74) | Placebo + Standard of Care. (N=76)
Hospitalization (Surgical and medical procedures) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Hospitalization (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion + Positively Smoke Free (N=72) | Bupropion + Standard of Care (N=72) | Placebo + Positively Smoke Free (N=74) | Placebo + Standard of Care. (N=76)
Dry Mouth (General disorders) | 21 (21) | 24 (24) | 34 (34) | 28 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2024-08-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT03342027/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2024-08-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT03342027/SAP_001.pdf